CLINICAL TRIAL: NCT05404698
Title: Integration of Multi-omics, Health Profile, Patient-related Outcomes and Exercise Data to Improve and Personalize Health Care in Hospital Settings: A CPExA Proof of Concept
Brief Title: Molecular and Clinical Response to a Single Bout of Aerobic Exercise in a Multimorbid Population: a Study From the Consortium on Precision EXercise in Aging
Acronym: CPExA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: Estrie University Integrated Health and Social Services Center - University Hospital of Sherbrooke (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-4591
Record Dates: First submitted 2022-05-18; First posted 2022-06-03 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-10

CONDITIONS: Multimorbidity - End-stage Kidney Disease
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Each participant performed 2 experimental conditions (rest, moderate continuous aerobic exercise with our cycle ergometer prototype - EXALT).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic intradialytic exercise (Experimental): 10 patients will perform Aerobic exercise with the cycle ergometer prototype (EXALT) during hemodialysis
  Interventions: Other: Aerobic exercise
- Standard care (Experimental): 10 patients will receive hemodialysis treatment (usual care)
  Interventions: Other: Control

INTERVENTIONS:
Other: Aerobic exercise — EX: 30 min of aerobic exercise (3/10 Borg scale) during hemodialysis treatment (between 30 min and 3h of treatment).
  Arms: Aerobic intradialytic exercise
Other: Control — CONT: participants will receive hemodialysis treatment only (usual care)
  Arms: Standard care

SUMMARY:
The combination of data from different origins (biological, health, patient-related) has the potential to improve care for the elderly. Precision approaches that are emerging in health are based on the premise that a better understanding of the biological responses to interventions will make it possible to optimize the treatments. In the field of exercise, this type of approach is emerging. This pilot study aims to collect preliminary data to demonstrate that a patient-centric vision with data from multiple sources is mandatory to personalize exercise intervention and improve health care. Older adults with end-stage chronic disease treated by hemodialysis represent a population of choice that requires personalized care since they are multimorbid and exhibit a complex health profile.

On the other hand, the beneficial effects of exercise are still little understood and the avoidance of adverse effects in response to exercise such as hypotension during dialysis remains uninvestigated.Objective: Demonstrate the feasibility of an integrative approach by combining "omics", clinical data, patient-related outcomes (PRO) as well as exercise variables (e.g., intensity, duration) Methods: A total of 10 people aged 60 and over will be recruited to randomly perform 2 experimental conditions: hemodialysis alone (CONT) or hemodialysis + aerobic exercise (EX), which will be carried out over 2 visits one week apart. These visits will take place at the scheduled time of the hemodialysis treatment. The variables of interest are: blood pressure response to a single bout of exercise exercise (during and post-exercise), symptoms (with visual analogue scales within 36 hours of the visit + Dialysis symptom index for the 7 days after the experimental visit), dialysis efficiency (Kt/V) and biological response (proteomics and metabolomics). Health-related quality of life (KDQOL questionnaire), medical data (electronic medical record), and level of physical activity (PASE questionnaire and smart watch; Apple Watch) will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* being treated by hemodialysis for end-stage kidney disease for at least 3 months
* medically eligible

Exclusion Criteria:

* diagnosed neurocognitive decline
* hip fracture with recent hemiarthroplasty preventing hip flexion while pedalling,
* COVID-19 positive,
* already included in another study.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-06-20 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
Change in blood pressure | Before and after the condition as well as every 5 minutes during the 20 minutes after (10 measurements). After this time frame, each 30 minutes up to the end of the dialysis session.
  Measured using standard clinical procedures (Automatic Blood Pressure Monitor at rest and with aneroid sphygmomanometer during and after exercise)
Change in perceived fatigue | Measured at 2:00 pm and 6:00 pm the day of the experimental condition and at 10:00 am, 2:00 pm and 6:00 pm the day following the experimental condition (for a total of 24 hours).
  10-centimeter horizontal visual analog scale, going from no fatigue (left) to extreme fatigue (right)
Change in perceived sleepiness | Measured at 2:00 pm and 6:00 pm the day of the experimental condition and at 10:00 am, 2:00 pm and 6:00 pm the day following the experimental condition (for a total of 24 hours).
  10-centimeter horizontal visual analog scale, going from no sleepiness (left) to extreme sleepiness (right)
Change in mood | Measured at 2:00 pm and 6:00 pm the day of the experimental condition and at 10:00 am, 2:00 pm and 6:00 pm the day following the experimental condition (for a total of 24 hours).
  10-centimeter horizontal visual analog scale, going from very bad (left) to very good (right)
Change in perceived soreness | Measured at 2:00 pm and 6:00 pm the day of the experimental condition and at 10:00 am, 2:00 pm and 6:00 pm the day following the experimental condition (for a total of 24 hours).
  10-centimeter horizontal visual analog scale, going from no soreness (left) to extreme soreness (right)
Change in perceived sleep quality | Measured at 10:00 am the day following the experimental condition.
  10-centimeter horizontal visual analog scale, going from very bad (left) to extreme soreness (right)
Plasma Metabolome and proteome at the end of the experimental (exercise) condition | After 30 minutes of exercise
  A blood draw will be realized immediately at the end of the dialysis session comprising the exercise condition. The plasma metabolome and proteome will be determined using mass spectrometry.
Plasma Metabolome and proteome at the end of the control (rest) condition | After 30 minutes of rest
  A blood draw will be realized immediately at the end of the dialysis session representing the control condition. The plasma metabolome and proteome will be determined using mass spectrometry.
Single pool Kt/V, experimental (exercise) condition | After 4 hours of dialysis
  measured using standard clinical procedures (blood draw before and at the end of the dialysis session comprising the exercise condition, by a research nurse).
Single pool Kt/V, control (rest) condition | After 4 hours of dialysis
  measured using standard clinical procedures (blood draw before and at the end of the dialysis session representing the condition, by a research nurse).

SECONDARY OUTCOMES:
Hematocrit (%) | Extracted from each patient's medical record at inclusion.
  Routinely measured (monthly) as standard clinical practice, before a dialysis session.
Hemoglobin (g/L) | Extracted from each patient's medical record at inclusion.
  Routinely measured (monthly) as standard clinical practice, before a dialysis session.
Red blood cells count (10^12/L) | Extracted from each patient's medical record at inclusion.
  Routinely measured (monthly) as standard clinical practice, before a dialysis session.
White blood cells count (10^9/L) | Extracted from each patient's medical record at inclusion.
  Routinely measured (monthly) as standard clinical practice, before a dialysis session.
Platelets count (10^9/L) | Extracted from each patient's medical record at inclusion.
  Routinely measured (monthly) as standard clinical practice, before a dialysis session.
Red blood cell mean corpuscular hemoglobin (pg) | Extracted from each patient's medical record at inclusion.
  Routinely measured (monthly) as standard clinical practice, before a dialysis session.
Red blood cell mean corpuscular volume (fL) | Extracted from each patient's medical record at inclusion.
  Routinely measured (monthly) as standard clinical practice, before a dialysis session.
Red blood cell distribution width (%) | Extracted from each patient's medical record at inclusion.
  Routinely measured (monthly) as standard clinical practice, before a dialysis session.
Plasma sodium (mmol/L) | Extracted from each patient's medical record at inclusion.
  Routinely measured (monthly) as standard clinical practice, before a dialysis session.
Plasma potassium (mmol/L) | Extracted from each patient's medical record at inclusion.
  Routinely measured (monthly) as standard clinical practice, before a dialysis session.
Plasma calcium (mmol/L) | Extracted from each patient's medical record at inclusion.
  Routinely measured (monthly) as standard clinical practice, before a dialysis session.
Plasma phosphate (mmol/L) | Extracted from each patient's medical record at inclusion.
  Routinely measured (monthly) as standard clinical practice, before a dialysis session.
Plasma glucose (mmol/L) | Extracted from each patient's medical record at inclusion.
  Routinely measured (monthly) as standard clinical practice, before a dialysis session.
Plasma creatinine (mmol/L) | Extracted from each patient's medical record at inclusion.
  Routinely measured (monthly) as standard clinical practice, before a dialysis session.
Health-Related Quality of Life | Once, at the beginning of the dialysis session comprising the first condition
  French version of the Kidney Disease Quality of Life 36 items version 1.3 (KDQOL-36)
Disease-related symptoms | Twice, seven days after each experimental conditions
  The French version of the Dialysis Symptom Index, consisting in a seven-day recall questionnaire assessing the presence and intensity of 30 symptoms
Physical activity scale for the Elderly (PASE) questionnaire | Once, at the beginning of the dialysis session comprising the first condition
  Recall questionnaire of the previous week's leisure, occupational and domestic physical activity habits validated in older adults.
Estimated daily energy expenditure | The watch will be worn during the 24 hours following each experimental condition
  Wrist-worn accelerometer (Apple Watch)

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Centre de recherche sur le vieillissement, Sherbrooke, Quebec
  - CIUSSS de l'Estrie - CHUS, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: No
Waiting for the University policy - standard operating procedures and data (upon ethics approval) would be available upon reasonable request